CLINICAL TRIAL: NCT03331484
Title: THE CAPITAL PCI AF Study: The Safety and Efficacy of Rivaroxaban and Ticagrelor for Patients With Atrial Fibrillation After Percutaneous Coronary Intervention
Brief Title: The Safety and Efficacy Of Rivaroxaban and Ticagrelor for Patients With Atrial Fibrillation After Percutaneous Coronary Intervention
Acronym: CAPITAL PCI AF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MRL-PCI AF
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation; Acute Coronary Syndrome
Keywords: percutaneous coronary intervention; bleeding; atrial fibrillation; Ticagrelor; Rivaroxaban
MeSH Terms: conditions — Atrial Fibrillation; Acute Coronary Syndrome; Hemorrhage | interventions — Ticagrelor; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ticagrelor and Rivaroxaban (Other): All participants will be prescribed ticagrelor 90 mg twice daily and rivaroxaban 15 mg once daily for a year.
  Interventions: Drug: Ticagrelor; Drug: Rivaroxaban

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 90 mg twice daily
Drug: Rivaroxaban — Rivaroxaban 15 mg once daily (10mg for patients with moderate renal impairment, creatinine clearance: 30-50 mL/min by the Cockcoft Gault method)

SUMMARY:
Currently, there is minimal data on the combination of rivaroxaban and ticagrelor in patients with atrial fibrillation (AF) managed with percutaneous coronary intervention (PCI). Furthermore, there exists significant controversy among physicians in the use of oral anticoagulants in conjunction with antiplatelet therapy in this population. The present recommendation is triple therapy (aspirin + clopidogrel + warfarin), which has been related to major bleeding complications. Previous studies have shown that ticagrelor has been proven to be more effective in reducing the rate of death, new heart attacks, or strokes than the previously recommended drug, clopidogrel, and studies have shown that less bleeding occurs with rivaroxaban than with warfarin. Therefore, it would be ideal to investigate the two potent drugs, ticagrelor and rivaroxaban, in combination in order to gain insight in the management of these high-risk patients.

The CAPITAL PCI AF study is a phase 3 Health Canada regulated interventional study involving the use of investigational drugs. It is a non-randomized, open-design study. The investigational team is studying the highly potent drug Ticagrelor, which is prescribed to participants receiving a stent placement, given in combination with Rivaroxaban, an oral anticoagulant recommended for patients with AF. The primary clinical endpoint is a safety outcome measuring bleeding complications in participants with AF treated within one year of the index PCI. The primary efficacy endpoint is measured by the clinical outcomes of death, stroke, non-central nervous system systemic embolism, myocardial infarction, and stent thrombosis within one year of the index PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has undergone a PCI with stent placement, plus
2. Documented non-valvular atrial fibrillation (AF)* within 1 year before screening, OR >1 year before screening if patient had been receiving oral anticoagulation (OAC)therapy for the atrial fibrillation for 3 months immediately before the index PCI.

   * AF is defined by its presence on an electrocardiogram (ECG), Holter monitor, or any device that provides a rhythm strip documenting paroxysmal, persistent or, permanent atrial fibrillation.

Atrial flutter can be included as "AF equivalent". The stroke risk in patients with atrial flutter is not much different from that in AF. Furthermore, many patients diagnosed with atrial flutter subsequently develop AF. Hence, current guidelines recommend that OAC should be used in patients with atrial flutter similar to that in patients with AF.

Non-valvular AF is defined as the absence of moderate to severe mitral stenosis or the presence of a mechanical valve as per 2016 ESC guidelines.

Exclusion Criteria:

1. Age <18 years old
2. Any condition that contraindicates anticoagulant therapy or would confer an unacceptable risk of bleeding, such as, but not limited to:

   i. active internal bleeding, ii. bleeding at a non-compressible site, iii. bleeding diathesis within 30 days of PCI, iv. baseline platelet count <90,000/μL, v. history of intracranial hemorrhage, vi. clinically significant gastrointestinal bleeding within 12 months of PCI, vii. baseline INR > 1.5 in patients not prescribed VKA, suggesting underlying coagulation disorder.
3. History of stroke
4. Cardiogenic shock at the time of screening
5. Ventricular arrhythmias refractory to treatment at the time of screening
6. Calculated CrCl <30 mL/min at the time of screening
7. Known significant liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis), or liver function test (LFT) abnormalities at screening: alanine transaminase (ALT) >5 times the upper limit of normal or ALT >3 times the upper limit of normal plus total bilirubin >2 times the upper limit of normal
8. Hemoglobin level <90 g/dL at screening
9. Any severe condition that would limit life expectancy to less than 12 months
10. Major surgery, biopsy of a parenchymal organ, or serious trauma within the past 30 days
11. Incomplete staged PCI procedure (once completion of the staged PCI has occurred, the final PCI may become the index event)
12. CABG planned
13. Transient AF caused by a reversible disorder (e.g. thyrotoxicosis, pulmonary embolism, recent surgery)
14. Any condition other than non-valvular AF requiring long-term anticoagulation with VKAs such as moderate to severe mitral valve stenosis, mechanical heart valves, deep vein thrombosis, pulmonary embolism, or left ventricular thrombus
15. Known allergies, hypersensitivity, or intolerance to rivaroxaban or ticagrelor
16. Pregnant or planning to become pregnant while enrolled in this study, or unwilling to employ an investigator-approved method of birth control
17. Participation in a study with another investigational device or drug < four weeks
18. Is receiving systemic treatment with strong inhibitors of both cytochrome P450 (CYP) 3A4 and p-glycoprotein (P-gp; eg, the azole-antimycotic ketoconazole and the HIV-protease inhibitor ritonavir). Treatment with fluconazole is allowed.
19. CHADS-VASC <1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Composite of TIMI Bleeds | 12 months
  Composite of TIMI Major Bleed, Minor Bleed, and Bleeding requiring medical attention

SECONDARY OUTCOMES:
The frequency of the individual components of the primary endpoint | 12 months
  Frequency of TIMI major, TIMI Minor, and TIMI bleeding requiring medical attention
The composite of multiple adverse cardiovascular events (MACE) | 12 months
  The composite of cardiovascular death and stroke events and its individual components
The frequency of stent thrombosis | 12 months
All-cause mortality | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel Le May, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No